CLINICAL TRIAL: NCT03065790
Title: Early FDG PET/CT Imaging as a Measure of Response in Patients With Non-Hodgkin Lymphoma on Lenalidomide
Status: Terminated | Type: Observational
Why Stopped: Adequate recruitment was not reached to continue the study.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 54416
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 2-Deoxy-2-[18F]fluoro-D-glucose (FDG) — 2-Deoxy-2-[18F]fluoro-D-glucose (FDG)

SUMMARY:
Adult patients with non-Hodgkin lymphoma who will be treated with lenalidomide will undergo FDG PET/CT scan as an early evaluation of response to therapy. Changes in FDG uptake will be correlated response and long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, at least 18 years of age
* History of histologically confirmed NHL as assessed per medical record review.
* At least one site of measurable disease (per RECIST 1.1) that is seen on CT, MRI, or FDG PET/CT.
* Recommended to start lenalidomide.
* Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Females who are pregnant or breast-feeding at the time of screening will not be eligible for this study. Female participants of child-bearing potential will have a urine or serum pregnancy test at the time of the screening visit.
* Inability to tolerate imaging procedures in the opinion of the investigator or treating physician.
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-Hodgkins Lymphoma
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Number of FDGmax SUV % change in FDG SUVmax | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farwell, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States